CLINICAL TRIAL: NCT02626663
Title: The Role of Microparticles as a Biomarker in Distinguishing Between Thrombotic Thrombocytopenic Purpura (TTP) and Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: The Role of Microparticles as a Biomarker
Status: Withdrawn | Type: Observational
Why Stopped: PI left the University, sponsor pulled funding
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Majed Refaai, Associate Professor, University of Rochester
Other Study IDs: RSRB00059370
Record Dates: First submitted 2015-10-20; First posted 2015-12-10 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Atypical Hemolytic Uremic Syndrome; Thrombotic Thrombocytopenic Purpura; Microparticles; Microangiopathic Hemolytic Anemia
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Purpura, Thrombotic Thrombocytopenic; Anemia, Hemolytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — platelet poor plasma samples will be retained. These samples will contain Microparticles and nanoparticles as well as microRNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- aHUS: atypical Hemolytic Uremic Syndrome
- TTP: Thrombotic thrombocytopenic purpura
- MAHA: other microangiopathic hemolytic anemias

SUMMARY:
The investigators propose to characterize MPs in aHUS and TTP both at the onset and throughout treatment. The investigators believe that the number, size, and cell origin of MPs will differ between these two diseases. The hypothesis is that endothelial derived MPs will be higher in number and comprise a larger portion of the MP population in aHUS and that platelet MPs will comprise a larger number and greater proportion of MPs in TTP. The investigators believe that MP identity and number can be used to reliably differentiate between aHUS and TTP at disease onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MAHA, TTP, and/or aHUS

Exclusion Criteria:

* Prisoners

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with Microangiopathic Hemolytic Anemias (MAHA), TTP, and/or aHUS are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Microparticle/Nanoparticle number (an absolute number) | an average of 3 months
Microparticle/Nanoparticle size (in nanometers or micrometers) | an average of 3 months
Microparticle/Nanoparticle identity (identity of cell type from which they are derived) | an average of 3 months

SECONDARY OUTCOMES:
Morbidities | 3 months
Mortality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schmidt, MD PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States